CLINICAL TRIAL: NCT05913713
Title: High Intensity Interval Training: Optimizing Exercise Therapy to Mitigate Cardiovascular Disease Risk Following Breast Cancer Chemotherapy
Brief Title: HIIT Following Breast Cancer Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB202300460 -N; 1R21AG078995-01A1 (NIH)
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training (HIIT) (Experimental): Supervised home-based high-intensity interval training will be performed on an all-extremity stationary cycle 3 days/week for 12 weeks.
  Interventions: Behavioral: 12-week Intervention Period; Behavioral: 12-week Observation Period
- Moderate Intensity Continuous Training (MICT) (Experimental): Supervised home-based moderate-intensity continuous training will be performed on an all-extremity stationary cycle 3 days/week for 12 weeks.
  Interventions: Behavioral: 12-week Intervention Period; Behavioral: 12-week Observation Period
- Usual Care (UC) (Other): Research participants will continue their habitual physical activity for the duration of the study. Once they complete the study, they will have the opportunity to perform supervised HIIT or MICT at home for 3 days/week for 12 weeks (research participants can choose either type of exercise).
  Interventions: Behavioral: 12-week Intervention Period; Behavioral: 12-week Observation Period

INTERVENTIONS:
Behavioral: 12-week Intervention Period — Research participants will be randomly assigned to either high-intensity interval training (HIIT), moderate-intensity continuous training (MICT), or the usual care (UC) group for a 12-week intervention period.
Behavioral: 12-week Observation Period — After a 12-week intervention period (HIIT, MICT, or UC), research participants will have a 12-week observation period to assess the durability of two types of different exercises.

SUMMARY:
Chemotherapy is an effective breast cancer treatment, which helped to increase the 5-year survival rate to approximately 95%. However, breast cancer survivors have a higher risk of cardiovascular disease (CVD) due to chemotherapy than adults without cancer. Cardiovascular rehabilitation can be an effective strategy to decrease the incidence of CVD and its risk factors in this population. The proposed study may help to examine the effect and durability of a novel high-intensity interval training compared to moderate-intensity continuous training on cardiovascular rehabilitation in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* female patients based on biological sex
* 18 to 85 years of age
* diagnosis of primary, invasive, non-metastatic, stages I-III breast cancer
* completed chemotherapy for breast cancer (anthracycline, alkylating agent and/or taxane) more than 6 months but less than 18 months prior to study enrollment. Adjuvant endocrine therapy for breast cancer (e.g., ovarian suppression, SERMs, SERDs, AIs), CDK4/6 inhibitors, PARP inhibitors, HER2 targeted agents, immunotherapy, and bisphosphonates are allowed within 6 months of study enrollment and during study participation
* absence of contraindications to exercise or to participate in study
* study clinician approval

Exclusion Criteria:

* do not meet inclusion criteria
* scheduled to receive surgery or radiation therapy during the intervention period
* any relevant cardiovascular diseases (stroke, heart failure, myocardial ischemia during maximal graded exercise test, myocardial infarction, angina pectoris, coronary artery bypass surgery or angioplasty or coronary stent)
* lymphedema stage ≥2 prior to study enrollment
* are pregnant
* current participation in other experimental interventions that may confound interpretation of study findings (e.g., dietary intervention for weight loss)

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who received chemotherapy for breast cancer
Enrollment: 158 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in brachial FMD | Baseline, Following a 12-week intervention period, Following a 12-week observation period
  Flow-mediated dilation (FMD) is an established non-invasive measure of endothelial function. Brachial artery FMD will be determined via ultrasonography in response to reactive hyperemia following 5-min forearm ischemia.
Change in cardiac function (global longitudinal strain) | Baseline, Following a 12-week intervention period, Following a 12-week observation period
  Global longitudinal strain is a marker of acute subclinical cardiotoxicity and is recommended for monitoring cancer patients at risk of cancer therapy-related cardiac dysfunction.
Percent completed vs. planned exercise frequency | Throughout the 12 weeks of supervised home-based exercise training
  The investigators will collect information throughout the exercise intervention regarding % completed vs. planned exercise sessions/week.
Percent completed vs. planned exercise duration | Throughout the 12 weeks of supervised home-based exercise training
  The investigators will collect information throughout the exercise intervention regarding % completed vs. planned exercise min/session.
Percent completed vs. planned exercise intensity | Throughout the 12 weeks of supervised home-based exercise training
  The investigators will collect information throughout the exercise intervention regarding % completed vs. planned exercise intensity/session.
Number of participants who experience adverse events as defined by most recent CTCAE throughout the exercise intervention | Throughout the 12 weeks of supervised home-based exercise training
  To evaluate safety plans are in place for determination and monitoring of adverse events according to the most recent National Cancer Institute Common Terminology Criteria for Adverse Events. Classification for seriousness, expectedness, severity and relationship to study intervention will be based on the NIH provided definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- Integrative Cardiovascular Physiology Laboratory, University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No